CLINICAL TRIAL: NCT05708027
Title: Two Strategies in Thoracoscopic Ablation for Lone Atrial Fibrillation
Brief Title: Thoracoscopic Ablation for Lone Atrial Fibrillation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal Research Clinical Center of Federal Medical & Biological Agency, Russia (Other Government)
Collaborators: Federal State Budget Institution Clinical Hospital, Moscow, Russia (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA-AF
Record Dates: First submitted 2022-10-26; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation; Heart Diseases
Keywords: Thoracoscopic ablation; Atrial Fibrillation; Ablation technique
MeSH Terms: conditions — Atrial Fibrillation; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AtriCure (Experimental): Group of patients to whom was applied AtriCure device during thoracoscopic ablation.
  Interventions: Procedure: Thoracoscopic surgical ablation
- Medtronic (Active Comparator): Group of patients to whom was applied Medtronic device during thoracoscopic ablation.
  Interventions: Procedure: Thoracoscopic surgical ablation

INTERVENTIONS:
Procedure: Thoracoscopic surgical ablation — Thoracoscopic surgical ablation is a minimally invasive procedure used to treat atrial fibrillation by creation Box Lesion Set using Radio Frequency Energy. Pulmonary veins isolation was performed using ablation clamps, whereas isolation of the posterior left atrium (box) was performed using a clamping Medtronic or a linear nonclamping AtriCure device.

SUMMARY:
Background: Thoracoscopic ablation is an effective treatment of patients with atrial fibrillation. Nowadays, 2 types of ablative devices are available in clinical practice allowing one to perform the thoracoscopic procedure - Medtronic and AtriCure. However, the contemporary clinical literature does not have enough data that would compare these two approaches.

Aims: to perform a comparative analysis of the short-term results of two minimally invasive strategies in thoracoscopic ablation for atrial fibrillation.

Methods:

The retrospective study was performed in which included 232 patients underwent thoracoscopic ablation for atrial fibrillation in two clinical centers for the period from 2016 to August 2021. The patients were divided into 2 groups. The first group was represented by those patients to whom a Medtronic device was applied (n=140), the second group was treated with an AtriCure device (n=92). The patients were comparable in their age, gender, initial severity of the condition. The follow-up consisted of laboratory tests, chest Х-ray, electrocardiography, 24-hour Holter monitor, echocardiography. The structure and prevalence of intraoperative and postoperative complications, specifics of the postoperative period were compared between the two groups.

DETAILED DESCRIPTION:
Patients of the thoracoscopic group were divided into 3 subgroups: I - low (no HF), II - medium (possible) and III - high risk of HF (HF confirmed) (Table 1). A statistically significant difference was found for the indicator: age (in the "high probability" group in relation to the "low probability" group by an average of 5.5 years; p=0.002) (Table 1). The clinical characteristics of patients in the studied subgroups are presented in Table 2, no significant difference was found for any of the compared indicators.

The nature of the cardiac arrhythmia and the severity of clinical symptoms are presented in Table 3. Significant differences were obtained for the following indicators: CHADS2VASc (in group III, "high probability" in relation to group I, "low probability" by an average of 1 point; p=0.008); HFA-PEFF (in group III, "high probability" by relative to group I "low probability" by an average of 5 points; p<0.001). Also, significant dynamics was obtained by the frequency of diagnosis of paroxysmal and long-lasting persistent forms of AF (p=0.025). Significant differences were obtained in the number of patients with 3 FC of heart failure (in group III, compared with group I, 5.3% vs 0.0%, respectively)

ELIGIBILITY:
Inclusion Criteria:

* persistent or long-lasting persistent form of atrial fibrillation;
* age over 18 years;
* failure of conservative therapy with the use of Class I and III antiarrhythmic drugs (Vaughan Williams classification);
* absence of marked structural pathology of the heart, requiring surgical treatment.

Exclusion Criteria:

* secondary atrial fibrillation due to reversible cause (pericarditis, hyperthyroidism, TELA, pneumonia, hypokalemia, etc.);
* surgical interventions on thoracic or mediastinal organs;
* age less than 18 years;
* presence of indications for open heart surgery under conditions of artificial circulation;
* heart failure with ejection fraction less than 30%;
* acute cerebral circulation disorder less than 3 months old;
* acute myocardial infarction or coronary stenting less than 3 months old;
* active systemic infection;
* left atrial appendage thrombosis detected one day before surgery;
* hemodynamically significant atherosclerotic lesion of coronary arteries and myocardial ischemia at the time of indications for surgery (confirmed by functional tests and coronarography);
* presence of contraindications for direct and indirect anticoagulants;
* presence of concomitant diseases of other organs and systems, which can lead to death within the first 2 years after the operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
The number of intraoperative complications | Day 1
  The number of intraoperative complications (Mortality, Stroke, Transient ischaemic attack, Sternotomy for bleeding, Mini-sternotomy for bleeding, Mini-thoracotomy for bleeding, Bleeding with discontinuation of procedure)
Postoperative complications | 1 mounth
  Postoperative complications: Major complications (Death, Reinterventions, Re-intubation without haemodynamic instability, Re-intubation due to haemodynamic instability, Venous lung infarction, Lung emboli, Permanent phrenic nerve paralysis, Stroke, Transient ischaemic attack, Atrium-oesophagus fistula, Myocardial infarction, Renal failure necessitating dialysis, Sepsis) and Minor complications (Pericardial fluid necessitating pericardiocentesis, Permanent pacemaker implantation, Thoracostomy drain, Infections, Delirium, Gastrointestinal bleeding)
Heart rhythm | at the time of discharge
  Heart rhythm (sinus rhythm, atrial fibrillation, pacemaker rhythm)

SECONDARY OUTCOMES:
Recurrence of atrial fibrillation | period after 3 month - 5 year.
  Development of recurrence of atrial fibrillation after thoracoscopic ablation
Cardiac Remodeling | after discharge - 5 year
  Assessment cardiac remodeling after thoracoscopic ablation (indexed left atrial volume, ejection fraction, systolic pulmonary artery pressure)
Functional class of heart failure | 1-5 year.
  Assessment of the functional class of heart failure after thoracoscopic ablation
Stroke and Transitory ischemic attack | after discharge - 5 year
  Development of Stroke and Transitory ischemic attack after thoracoscopic ablation
Unplanned cardiovascular hospitalization | after discharge - 5 year
  Unplanned non-cardiovascular hospitalization after thoracoscopic ablation

CONTACTS AND LOCATIONS:
Overall Officials: Alexander V Troitskiy, MD, SD, Study Director — Federal Research and Clinical Center
Locations (2):
- Russia (2):
  - Federal State Budget Institution Clinical hospital, Moscow
  - Federal Research Clinical Center of Federal Medical & Biological Agency, Moscow

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data (IPD).

REFERENCES:
- [Background] Zotov AS, Troitsky AV, Silaev AA, Sakharov ER, Sukhotin VN, Shelest OO, Khabazov RI, Timashkov DA. Short-Term Results of Two Strategies in Thoracoscopic Ablation for Lone Atrial Fibrillation. Journal of Clinical Practice. 2022;13(3):5-16.doi: https://doi.org/10.17816/clinpract110719